CLINICAL TRIAL: NCT04845425
Title: Identification of miRNAs in Endometrial Cancer as Novel Diagnostic and Prognostic Biomarkers
Brief Title: Analysis of miRNA Expression in Endometrial Cancer
Acronym: MIRCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Anna Myriam Perrone, Principal investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: 189/2021/Oss/AOUBo
Record Dates: First submitted 2021-04-10; First posted 2021-04-15 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; miRNA; microRNA; TGCA
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The TCGA project identified four distinct prognostic groups of endometrial carcinoma (EC) based on molecular alterations: (i) the ultramutated subtype that encompasses POLE mutated (POLE) cases; (ii) the hypermutated subtype, characterized by MisMatch Repair deficiency (MMRd); (iii) the copy-number high subtype, with p53 abnormal/mutated features (p53abn); (iv) the copy-number low subtype, known as No Specific Molecular Profile (NSMP). Although the prognostic value of TCGA molecular classification, NSMP carcinomas present a wide variability in molecular alterations and biological aggressiveness. Given that the study aims to evaluate the miRNA expression profile to identify novel potential biomarkers to better stratify the EC patients, taking into account the molecular status

ELIGIBILITY:
Inclusion Criteria:

* age>18yo
* histological diagnosis of endometrial cancer
* tumor resection
* patient's informed consent

Exclusion Criteria:

* patients with other neoplasia within the last 5 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with endometrial cancer
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of miRNA expression based on the 4 molecular groups | 1 year
  Evaluate miRNA expression based on the 4 molecular groups recently identified

SECONDARY OUTCOMES:
Integration of molecular results with clinico-pathological data | 1 year
  Integration of molecular results with clinico-pathological data

CONTACTS AND LOCATIONS:
Overall Officials: Anna Myriam Perrone, Principal Investigator — IRCCS Azienda Ospedaliera-Universitaria di Bologna
Locations (1):
- IRCCS- Azienda Ospedaliera-Universitaria di Bologna, Bologna, Bo, Italy

IPD SHARING:
Plan to Share IPD: No